CLINICAL TRIAL: NCT03846011
Title: Metabolic Evaluation of Urolithiasis: Comparison of 24-hour Collecting Urine Prior and After Stone Removal - a Prospective Study
Brief Title: Comparison of 24-hour Collecting Urine Prior and After Stone Removal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Head of the department of urology, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 2019-003
Record Dates: First submitted 2019-01-26; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Urolithiasis; Urinary Stone
Keywords: urolithiasis; 24-h urine composition
MeSH Terms: conditions — Urolithiasis; Urinary Calculi | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experiment group: All eligible patients administered for active stone removal.
  Interventions: Other: 24-h urine collection

INTERVENTIONS:
Other: 24-h urine collection — Collecting 24-h urine prior and after stone removal surgery

SUMMARY:
The metabolic evaluation is crucial for determining possible underlying diseases causing stone growth and to consider the lifestyle changes or medical prophylaxis needed to prevent or at least reduce stone recurrence. 24-hour urine collection is the main part of the metabolic evaluation. The time point is suggested between 3 weeks and 3 month after stone removal, but so far there are no studies comparing 24-hour urine prior and after stone removal. In this study, investigators would like to analyze parameters in the 24-hour urine prior and after complete stone removal to see whether metabolic status can be evaluated no matter stone free or not.

DETAILED DESCRIPTION:
Background As the metabolic evaluation is an essential part of diagnostic and recurrence prevention of urolithiasis, the current EAU Guidelines, as well as the German S2k guidelines therefore suggest 24-hour urine collection, done twice. This evaluation is crucial for determining possible underlying diseases causing stone growth and to consider the lifestyle changes or medical prophylaxis needed to prevent or at least reduce stone recurrence.

The time point is suggested between 3 weeks and 3 month after stone removal, but so far there are no studies comparing 24-hour urine prior and after stone removal. This could simplify the diagnostic and make this essential information available for more patients suffering from urolithiasis.

Hypothesis

Null hypothesis: The analyzed parameters in the 24-hour urine prior and after complete stone removal differ from each other Alternative hypothesis: The analyzed parameters in the 24-hour urine prior and after complete stone removal do not differ from each other Primary endpoint: The difference of the analyzed parameters prior and after complete stone removal

Parameters to be collected

1. 24h urine composition prior and after stone removal: pH value, spec. weight, creatinine, calcium, oxalate, uric acid, citrate, magnesium, phosphate, ammonium, cysteine, sodium, potassium.
2. Secondary: Age, sex, body mass index, stone composition analyzed by infrared spectroscopy, urine culture, comorbidities (diabetes mellitus, hypertension, …), degree of hydronephrosis, serum electrolytes, blood urea nitrogen, serum creatinine, first manifestation or recurrent disease

Methods

* After assessing inclusion and exclusion criteria, all eligible patients administered for active stone removal are included in this study.
* Prior to surgery, a 24-hour urine collection need to be performed (not longer than 2 month).
* Post-operatively stone free status is assessed by NCCT, in ureterolithiasis only if stone free status is uncertain.
* 4 weeks after proven stone free status the post surgical 24h urine collection is performed.
* If a ureter stent was placed, the 24-hour urine collection is performed 4 weeks after stent removal.
* All 24-hour collection are performed as outpatients. Patients will be asked to drink and eat normally when they do their urine collection. Urinary volume is measured as a marker of liquid consumption, sodium as a marker of salt intake.

Sample size As no available data to show the difference of urine composition prior or after surgery, the study will enroll 100 participants first to get preliminary data. Then the final sample size will be determined by the preliminary data.

Statistical Analysis： Comparisons of the urine compositions before and after stone removal will be performed using the Student's t-test for continuous variables and chi-squared for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Urolithiasis (Nephrolithiasis, Ureterolithiasis)

Exclusion Criteria:

* Patients under 18 years
* Urinary tract infection (positive urine culture prior to surgery)
* Incomplete 24h urine collection
* Pregnancy
* Residual stones after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urolithiasis patients administered for active stone removal
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Urine pH Change | Change from baseline urine pH at 4 weeks after proven stone free status
  pH values will be determined with a glass electrode in a calibrated pH meter
24-h Urine oxalate excretion change | Change from baseline 24-h urine oxalate excretion at 4 weeks after proven stone free status
  Urine oxalate will be measured using ion exchange chromatography
24-h Urine citrate excretion change | Change from baseline 24-h urine citrate excretion at 4 weeks after proven stone free status
  Urine citrate will be measured using ion exchange chromatography
24-h Urine calcium excretion change | Change from baseline 24-h urine calcium excretion at 4 weeks after proven stone free status
  Urine calcium will be measured by Unicel DxC 600 synchronic biochemical detecting system.
24-h Urine phosphate excretion change | Change from baseline 24-h urine phosphate excretion at 4 weeks after proven stone free status
  Urine phosphate will be measured by Unicel DxC 600 synchronic biochemical detecting system.
24-h Urine sodium excretion change | Change from baseline 24-h urine sodium excretion at 4 weeks after proven stone free status
  Urine sodium will be measured by Unicel DxC 600 synchronic biochemical detecting system.
24-h Urine potassium excretion change | Change from baseline 24-h urine potassium excretion at 4 weeks after proven stone free status
  Urine potassium will be measured by Unicel DxC 600 synchronic biochemical detecting system.
24-h Urine chloride excretion change | Change from baseline 24-h urine chloride excretion at 4 weeks after proven stone free status
  Urine chloride will be measured by Unicel DxC 600 synchronic biochemical detecting system.
24-h Urine creatinine excretion change | Change from baseline 24-h urine creatinine excretion at 4 weeks after proven stone free status
  Urine creatinine will be measured by Unicel DxC 600 synchronic biochemical detecting system.
24-h Urine uric acid excretion change | Change from baseline 24-h urine uric acid excretion at 4 weeks after proven stone free status
  Urine uric acid will be measured using Beckman coulter AU680 automatic biochemistry analyzer.
24-h Urine magnesium excretion change | Change from baseline 24-h urine magnesium excretion at 4 weeks after proven stone free status
  Urine magnesium will be measured using Beckman coulter AU680 automatic biochemistry analyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu W, Zhang X, Lu S, Ozsoy M, Zhou Z, Huang Z, Ai G, Zeng G. Comparison of 24-hour urine composition prior to and after stone removal in nephrolithiasis: a prospective observational study. Minerva Urol Nephrol. 2024 Jun;76(3):351-356. doi: 10.23736/S2724-6051.22.05164-3. Epub 2023 Feb 13. PMID 36779823